CLINICAL TRIAL: NCT06471608
Title: Impact of Ambulatory Management for Primary Spontaneous Pneumothorax in the Emergency Department on Quality of Life: a Randomized Clinical Trial
Brief Title: Impact of Ambulatory Management for Primary Spontaneous Pneumothorax in the Emergency Department on Quality of Life
Acronym: EFFI-PNO
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 9155
Record Dates: First submitted 2024-06-14; First posted 2024-06-24 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: Primary Spontaneous Pneumothorax; Quality of Life; Ambulatory Care; Chest Tube
Keywords: Chest tube drainage; Primary spontaneous pneumothorax; Ambulatory management; Quality of life
MeSH Terms: conditions — Pneumothorax | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard care (Active Comparator): Chest tube drainage with hospital management
  * chest tube drainage (with a straight or pigtail drain, less than ≤ 14 Fr in diameter, inserted using the Seldinger versus Seldinger technique, or using the standard drainage technique with an internal mandrel drain), followed by post-procedure imaging prior to transfer to the department, in accordance with standard practice (chest X-ray or low-dose CT scan, depending on management practices at the center).
  * Hospitalisation in a hospital department (pulmonology, thoracic surgery, short-stay emergency unit, critical care, according to the usual pathway of the center in which the patient is included).
  * In-hospital monitoring until complete resolution of pneumothorax and drain removal (average 4-6 days).
  Interventions: Other: Standard Care
- Ambulatory management (Experimental): - Chest tube drainage in emergency department (Furhmann drain connected to Heimlich valve), connected to suction system at -5 to -10 cm H2O until bubbling stops and ambulatory management after monitoring in the emergency department
  Interventions: Other: Ambulatory management

INTERVENTIONS:
Other: Ambulatory management — * Chest tube drainage in emergency department (Furhmann drain connected to Heimlich valve), connected to suction system at -5 to -10 cm H2O until bubbling stops
  * Follow-up imaging at 4 hours (chest X-ray or low-dose CT scan, depending on management practices in the centers)
    * if the pneumothorax is still very large, or if clinical tolerance is unsatisfactory (dyspnea, unrelieved pain, abnormal vital parameters), the patient should be admitted to hospital
    * if the lung is in the process of reattachment and a minimal detachment persists, and clinical tolerance is good (assessed on vital parameters, with oxygen saturation above 98%, good hemodynamic stability and pain relieved by analgesics), the patient may be discharged home.
  Arms: Ambulatory management
Other: Standard Care — Hospitalisation in a hospital department (pulmonology, thoracic surgery, short-stay emergency unit, critical care, according to the usual pathway of the center in which the patient is included).
  In-hospital monitoring until complete resolution of pneumothorax and drain removal (average 4-6 days).
  Arms: Standard care

SUMMARY:
Outpatient treatment of Primary Spontaneous Pneumothorax (PSP) compared to usual inpatient management could improve quality of care and represent a more efficient, generalizable and sustainable strategy.

This multicenter, cluster-controlled, randomized interventional study with stepped wedge implementation will evaluate the impact on quality of life (between inclusion, after drain placement, and 6 months) of an ambulatory strategy for the management of large abundance primary spontaneous pneumothorax in the emergency department, compared with usual care.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 to 50 years presenting to the emergency department with a 1st episode of right or left primary spontaneous pneumothorax (PSP) of large abundance diagnosed by chest X-ray or CT scan defined according to British Thoracic Society (BTS) recommendations as a detachment greater than 2 cm over the entire height of the axillary line.
* Patient living less than an hour from hospital and able to be accompanied for the first 48 hours
* Patient able to understand the aims and risks of the research and to give informed, dated and signed consent
* Patient with Internet access and able to complete online questionnaires
* Patient affiliated to or benefiting from a social health insurance

Exclusion Criteria:

* Small pneumothorax (≤ 2cm)
* Suffocating pneumothorax defined by the presence of signs of respiratory distress or hemodynamic failure with indication for emergency exsufflation
* Patient on emergency oxygen or long-term oxygen therapy
* Traumatic pneumothorax
* Secondary spontaneous pneumothorax
* Bilateral pneumothorax
* Associated fluid effusion
* Risk-benefit balance unfavorable to outpatient treatment (comorbidities, isolated patient, difficulty understanding monitoring instructions)
* Patient living more than one hour from hospital
* Patients living alone or unable to be accompanied on discharge for the first 48 hours
* Patients under legal protection
* Pregnant or breast-feeding women
* Patient participating in a therapeutic interventional clinical trial or in a period of exclusion linked to previous participation in a clinical trial

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 386 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2030-07-01 (Estimated); Study Completion 2030-07 (Estimated)

PRIMARY OUTCOMES:
Quality of life at 6 months | 6 months
  Evaluate the impact on quality of life (between inclusion, after drain placement, and 6 months) of an ambulatory strategy for the management of large abundance primary spontaneous pneumothorax in the emergency department, compared with usual care, using the Short Form (36) Health Survey (The lower the score the more disability)

SECONDARY OUTCOMES:
Success rate of the strategy as measured by pulmonary expansion (lung reattachment on X-ray / CT scan) the latest by the investigator who performed the drainage procedure | Day 6
Proportion of patients having benefited from an exclusive outpatient management (patients not requiring hospitalisation during the ambulatory approach) | Day 6
Assessment of Pain | Day 0, Day 2, Day 4, Day 6 and monthly
  Pain assessed on a numerical scale (rated from 0 to 10), 0 being the lowest pain and 10 being the maximum pain
Assessment of Dyspnea according to the mMRC classification | Day 0, Day 2, Day 4, Day 6 and monthly
  mMRC classification (0 to 4), 0 being no discomfort and 4 shortness of breath for simple acts of daily living.
Complication rates (major and minor) in the 2 groups | Day 2, 4, 6, 1 month and 1 year
  * Minor (bleeding at insertion site, tube kinking, pain limiting inspiratory movements, subcutaneous emphysema, unsightly scar)
  * Major (hemothorax due to lesion of the vasculonervous bundle, bubbling (leakage) at the tube insertion site, accidental removal, perforation of an organ (lung, spleen, etc.), local abscess, iatrogenic pneumothorax on tube removal, pulmonary re-expansion edema).
Pneumothorax Recurrence Rate | at 1 year
  Incidence of recurrence in both groups.
Patient satisfaction assessed by SAPS (The Short Assessment of Patient Satisfaction) questionnaire | Day 0, 1 month, 6 months and 1 year
Patient preference (coded from 0 to 5): ambulatory/non-ambulatory | Day 0, 1 month, 6 months and 1 year
  Preference will be assessed as follows: Each patient will be asked to code their opinion of outpatient management from 0 to 5, and their opinion of inpatient management from 0 to 5, whatever their randomization group (0 being the worst opinion of the strategy, and 5 a very positive opinion of the strategy).
Anxiety assessed by the State-Trait Anxiety Inventory (STAI) | Day 0, 1 month, 6 months and 1 year.
Quality of life assessed by SF-36 (The Short Form (36) Health Survey) | at 1 month and 1 year
Ambulatory strategy implementation criteria : Penetrance | At 1 year
  Assesses how widely the device is deployed within a service and whether it is transferable to other contexts. Studied through focus groups with professionals on adoption, institutional changes, and scalability
Ambulatory strategy implementation criteria : Acceptability | At 1 year
  Represents how patients and healthcare professionals perceive the benefits and limits of the device in care and relationships. Evaluated through semi-structured interviews (patients' experiences) and focus groups (care practices)
Ambulatory strategy implementation criteria : Appropriation | At 1 year
  Concerns the perceived added value of the device in care management and patient-professional relations. Measured via interviews (perceived value/efficacy) and focus groups (use in ambulatory vs hospital care).
Ambulatory strategy implementation criteria : Adoption | At 1 year
  Refers to whether professionals and patients integrate or learn new practices with the device. Assessed by interviews on experiences and focus groups on care practices.
Ambulatory strategy implementation criteria : Feasibility | At 1 year
  Looks at the practical experience of using the device in daily care and the caregiver-patient relationship. Explored in focus groups with healthcare professionals discussing usability and practicality.
Ambulatory strategy implementation criteria : Fidelity | At 1 year
  Examines whether the device is applied as initially intended, and the perceived quality of its implementation. Assessed through focus groups reflecting on adherence to goals and strategies in care delivery.
Ambulatory strategy implementation criteria : Cost of implementation | At 1 year
  Considers the economic impact for patients and the health system (direct and indirect costs). Evaluated through quantitative patient data: hospital stays, readmissions, and insurance compensation.
Ambulatory strategy implementation criteria : Durability | At 1 year
  Relates to maintaining the device over time and integrating it into routine care across hospitals. Evaluated via interviews (patients' risk perception, care continuity) and focus groups (staff reflection on long-term use).
Duration of emergency care in the 2 groups | 1 year
Estimation of costs associated with each strategy | at 1 year
  Total direct and indirect healthcare costs associated with each management strategy.
Estimation of the difference in QALYs gained using a mixed model | at 1 year
Incremental cost-utility ratio, defined as the difference in costs divided by the difference in utility estimated by the EQ-5D scores obtained by mapping from the SF-36 | at 1 year
  with a valuation of the scores obtained with the utilities published for the French population
Budgetary impact of a national roll-out scenario for the ambulatory care strategy from the perspective of the French Health Insurance | at 1 year

CONTACTS AND LOCATIONS:
Locations (7):
- France (7):
  - CHRU de Besançon - Hôpital Jean Minjoz, Besançon
  - Hôpital Pellegrin - CHU de Bordeaux, Bordeaux
  - CHU de Grenoble - Hôpital Michallon, La Tronche
  - Hôpital Saint Louis - AP-HP, Paris
  - Hôpital Universitaire Pitié Salpétrière AP-HP, Paris
  - Hôpital de la Milétrie - CHU de Poitiers, Poitiers
  - Hôpitaux Universitaires de Strasbourg, Strasbourg

REFERENCES:
- [Derived] Kepka S, Wilme V, Duracinsky M, Matau C, Nze Ossima A, Gil Jardine C, Le Borgne P, Marjanovic N, Marx T, Ohana M, Peyrony O, Philippon AL, Viglino D, Chenou A, Clere-Jehl R, Bilbault P, Durand-Zaleski I, Sauleau EA. Ambulatory management of primary spontaneous pneumothorax in the emergency department: EFFI-PNO protocol - a multicentre, cluster-controlled, stepped-wedge, randomised interventional study. BMJ Open. 2025 Dec 24;15(12):e106739. doi: 10.1136/bmjopen-2025-106739. PMID 41448686